CLINICAL TRIAL: NCT04163848
Title: CARbon Impact of aNesthesic Gas - A Carbon Footprint Comparison of Sevoflurane and Desflurane in an Optimized Fresh Gas Flow Protocol
Brief Title: CARbon Impact of aNesthesic Gas
Acronym: CARING
Status: Completed | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Olivier Verdonck, Assistant Professor, Deputy chief of the Department of Anesthesiology of Maisonneuve-Rosemont Hospital, University of Montreal(UDeM), Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 2020-1971
Record Dates: First submitted 2019-11-06; First posted 2019-11-15 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Gas; Inhalation; Anesthesia
Keywords: Desflurane; Sevoflurane; Fresh gas flow; Environment
MeSH Terms: conditions — Mucopolysaccharidosis IV; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Desflurane: desflurane administration based on a BIS index kept between 40-60 and with use of the semi-closed circuit of the Draeger A500 ventilator and its econometer for an optimized fresh gas flow as low as the O2 consumption allows
  Interventions: Other: Pollution
- Sevoflurane: sevoflurane administration based on a BIS kept between 40-60 and with use of the semi-closed circuit of the Draeger A500 ventilator with a fixed fresh gas flow of 2L/min as requested in the gas monography
  Interventions: Other: Pollution

INTERVENTIONS:
Other: Pollution — CO2 equivalent productions related to anesthetic gases use during general anesthesia for laparoscopic surgery

SUMMARY:
Assessing the impact of anesthesia practice on global warming and carbon footprint becomes part of the standard of care and is growing concern within the anesthesia community. Global Warming Potential (GWP) is a measure of how much a given mass of greenhouse gas contributes to global warming over a specified time period. Inhaled anesthetics have various GWP20: 349 for sevoflurane and 3714 for desflurane. However, GWP20 and CDE20 alone are not sufficient to evaluate the environmental impact of anesthetic gases. Other parameters must be included in the analysis: fresh gas flow (FGF), carrier gas (air, O2, N2O) and potency of the anesthetic gas. Unfortunately, the majority of trials did not fully consider the FGF reduction and the fact that desflurane can be administered with new closed or very low-flow anesthesia circuits as opposed as the recommended 2L/min that must be used for sevoflurane according to its monography in Canada. Most of the calculations were made on a purely theoretical approach that could be different from actual measurements based on a strictly monitored anesthesia practice. When continuous and accurate gas monitoring and analysis is used as recommended nowadays, the use of closed or semi-closed-circuit anesthesia with very low FGF might allow for a reduction of more than 80% of the anesthetic gas administration and its consequent pollution. By properly monitoring the anesthesia depth and analgesia adequacy, the investigators can reduce the gas consumption. The proposed study will aim at determining whether with the help of high-quality monitoring (BIS and NOL) and high-end ventilators that allow minimal fresh gas flow, the use of desflurane remains more polluting than sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients,
* laparoscopic general, gynecological or urologic surgery requiring general anesthesia without additional regional anesthesia technique
* fully consented,
* BMI < 40,
* age > 18yo,

Exclusion Criteria:

* post-operative need for a neuraxial or regional analgesic technique
* history of active coronary artery disease
* serious cardiac arrhythmia (including atrial fibrillation)
* history of substance abuse
* chronic use of psychotropic and/or opioid drugs
* history of psychiatric diseases with the need of medication
* history of refractory PONV
* allergy or contra-indication to any drug used in the study protocol
* refusal of the patient for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population undergoing laparoscopic gynecologic, urologic or general surgery
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
CO2 equivalent of volatile inhaled anesthesic gases use in grams | From intubation to end of surgery
  To compare total volatile inhaled anesthetics consumption in CO2 equivalent (grams) per hour during anesthesia for laparoscopic surgery between two groups: Group "D" for Desflurane and group "S" for Sevoflurane

SECONDARY OUTCOMES:
Total volatile inhalated anesthesics consumption in mL | From intubation to end of surgery
  To compare the total volatile inhaled anesthetics consumption in mL, mL/h and mL/kg/h during anesthesia for laparoscopic surgery between desflurane and sevoflurane
Cost in dollars | From intubation to end of surgery
  To compare the total cost of volatile inhalated anesthesics (mL of gaz x $/mL of gaz) for each group
Extubation time in minutes | From stopping anesthesics gases to extubation
  To compare the extubation time
Recovery room time in minutes | From end of surgery to 240minutes post-surgery
  To compare the time spent in the recovery room

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Maisonneuve-Rosemont, CIUSSS de l'Est de l'Ile de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No